CLINICAL TRIAL: NCT01964443
Title: EPidemiological Study In Patients With Recently DiagnosEd PSOriasis: Clinical Assessment and Psychosocial Impact of This Disease
Brief Title: Clinical Assessment and Psychosocial Impact of Psoriasis
Acronym: EPIDEPSO
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100972; CNTO1275PSO4034 (Other: Janssen Pharmaceutica NV - CTMS ID)
Record Dates: First submitted 2013-09-17; First posted 2013-10-17 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Alexithymia; Quality of life
MeSH Terms: conditions — Psoriasis; Affective Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all included patients: Men and women, 18 years of age and older, who have had the onset of the first symptoms of plaque psoriasis less than 10 years before study entry, are naïve or experienced to topical treatment, and are eligible for phototherapy or systemic treatment

SUMMARY:
The purpose of this study is to explore the impact of plaque psoriasis on the different dimensions of patient life including psychological disorders, different types of addictions, and their consequences on health-related quality of life and socioeconomic parameters at baseline (cross-sectional part) and during the initial years of the psoriasis disease (longitudinal part).

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational, multicenter study to document the prevalence of alexithymia in adult men and women, 18 years of age and older, who have had the onset of the first symptoms of plaque psoriasis less than 10 years before study entry, are naïve or experienced to topical treatment, and are eligible for phototherapy or systemic treatment. Only data available from routine clinical practice will be collected and all treatment decisions will be made at the discretion of the treating physician. Additionally, where local regulations permit, participating physicians will be asked to obtain Patient-Reported Outcome (PRO) data from patients participating in this observational study. A target of 800 adult patients will participate in this study at approximately 80 sites. The enrollment period of this study is expected to continue for approximately 9 months. Each patient will receive treatment as per standard clinical practice and will be followed up for 12 months. Therefore, the total duration of this observational study is expected to be approximately 21 months. Overall psoriasis disease severity as assessed by the physician will be documented at baseline (cross-sectional) and in the observational (longitudinal) phase of the study. Several outcomes related to psychosocial comorbidities (eg, alexithymia, anxiety, depression), addiction, and work and activity impairment as measured by PRO questionnaires and scales will also be collected. Information on psoriasis treatment(s) (topical, phototherapy, systemic [non-biologic, biologic]), mental health drugs (including those used for sleep), and concomitant medications given for comorbid medical conditions will also be collected. The data for this study will be analyzed and reported separately for the cross-sectional data (baseline) and for the longitudinal data (from baseline to Month 12).

ELIGIBILITY:
Inclusion Criteria:

Have onset of first symptoms of plaque psoriasis less than 10 years before baseline; Be either naïve or experienced to topical treatment; Be eligible for phototherapy or systemic treatment, as determined by the participating physician at the patient's baseline visit.

Exclusion Criteria:

Has a history of or current treatment with a systemic agent (including biologic agents); Has non-plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular); Has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before the start of the study or first data collection time point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, 18 years of age and older, who have had the onset of the first symptoms of plaque psoriasis less than 10 years before study entry, are naïve or experienced to topical treatment, and are eligible for phototherapy or systemic treatment
Sampling Method: Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
prevalence of alexithymia | Baseline
  presence of alexithymia defined as 20-item Toronto Alexithymia Scale (TAS-20) score ≥61: TAS-20 is a validated self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale: 1 = strongly disagree, 2 = neither agree or disagree, 3 = undecided, 4 = agree, 5 = strongly agree. There are 3 subscales: difficulty describing feelings, difficulty identifying feelings, and externally oriented thinking. The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.

SECONDARY OUTCOMES:
psoriasis disease duration | baseline, month 6 and month 12
  Psoriasis Global Assessment (PGA): Overall lesions are graded for induration (from 0 = no evidence of plaque elevation to 5 = severe plaque elevation = 1.25 mm or more), erythema (from 0 = no evidence of erythema, hyperpigmentation may be present to 5 = dusky to deep red coloration), and scaling (from 0 = no evidence of scaling to 5 = severe; very thick tenacious scale predominates). The sum of the 3 scales is divided by 3 and rounded to obtain a final PGA score. The PGA final scores are defined as: 0 = cleared, except for residual discoloration; 1 = minimal; 2 = mild; 3 = moderate; 4 = marked; and 5 = severe.
psoriasis disease severity | baseline, month 6 and month 12
  Psoriasis Area and Severity Index (PASI): system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72. A PASI 50 response is defined as ≥50% improvement in PASI score from baseline; PASI 75 and PASI 90 are similarly defined.
anxiety and depression | baseline, month 6 and month 12
  Hospital Anxiety and Depression Scale (HADS; subscales: anxiety [-A], depression [-D]) is a validated 14-item scale with 7 of the items relating to anxiety and 7 relating to depression. Each item is scored from 0 to 3, with higher scores indicating greater likelihood of depression or anxiety. Cases of anxiety or depression are each defined by subscale scores of 8 or greater, and categorized as normal (score of 0 to 7), mild (score of 8 to 10), moderate (score of 11 to 14), and severe (score of 15 to 21). The recall period is the past week.
problematic drinking | baseline, month 6 and month 12
  Alcohol Use Disorders Identification Test (AUDIT) consists of 10 questions about a patient's quantity and frequency of alcohol use. The response to 8 of the questions are scored as 0 = never, 1 = monthly or less, 2 = 2 to 4 times a month, 3 = 2 to 3 times a week, 4 = 4 or more times a week. Two questions are scored as 0 = no, 2 = yes, but not in the last year, 4 = yes, during the last year. A score of 8 or more is associated with harmful or hazardous drinking. In this study, the patient self-report questionnaire will be used
smoking | baseline, month 6 and month 12
  number of cigarettes smoked per day
physical and mental/emotional quality of life | baseline, month 6 and month 12
  Dermatology Life Quality Index (DLQI) is a dermatology-specific validated 10-question quality of life instrument. Each question addresses how much the patient's skin problem has affected their life and is scored as: 3 = very much, 2 = a lot, 1 = a little, 0 = not at all, or 0 = not relevant. The recall period is the past week. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more health-related quality of life is impaired: 0 to 1 = no effect at all on patient's life; 2 to 5 = small effect on patient's life; 6 to 10 = moderate effect on patient's life; 11 to 20 = very large effect on patient's life; 21 to 30 = extremely large effect on patient's life.
work and activity impairment related to psoriasis | baseline, month 6 and month 12
  Work Productivity and Activity Impairment questionnaire:Psoriasis (WPAI:PSO) produces 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI:PSO outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, ie, worse outcomes.
alexithymia prevalence rate | month 6 and month 12

CONTACTS AND LOCATIONS:
Locations (48):
- Austria (2):
  - Graz
  - Vienna
- Belgium (4):
  - Edegem
  - Ghent
  - Liège
  - Mons
- France (8):
  - Brest
  - Martigues
  - Nice
  - Pierre-Bénite
  - Reims
  - Rouen
  - Toulouse
  - Vandœuvre-lès-Nancy
- Greece (4):
  - Athens
  - Heraklion
  - Thessaloniki
  - Thessalonikis
- Ireland (2):
  - Dublin
  - Galway
- Israel (6):
  - Afula
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Netherlands (4):
  - Alkmaar
  - Amsterdam
  - Breda
  - Nijmegen
- Norway (2):
  - Bergen
  - Tromsø
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- South Africa (2):
  - Bloemfontein
  - Durban
- Spain (7):
  - Albacete
  - Alcorcón
  - Alicante
  - Barcelona
  - Bilbao Vizcaya
  - Santander
  - Valencia
- United Kingdom (4):
  - Cardiff
  - Dundee
  - London
  - Salford